CLINICAL TRIAL: NCT05026658
Title: A Prospective, Randomized, Controlled Clinical Study to Evaluate the Agreement and Reproducibility of Visibly Digital Acuity Product
Brief Title: Prospective, Randomized, Controlled Agreement and Reproducibility Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Visibly (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: VDAP-1002
Record Dates: First submitted 2021-08-17; First posted 2021-08-30 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Digital Acuity Product

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Visibly Digital Acuity Product (Experimental)
  Interventions: Device: Visibly Digital Acuity Product
- ETDRS Visual Acuity Lane Test (Experimental)
  Interventions: Device: Visibly Digital Acuity Product

INTERVENTIONS:
Device: Visibly Digital Acuity Product — The order of testing (two VDAP home environments and ETDRS) will be randomly assigned for each subject as one of four sequences:
  1. V1, E, V2
  2. E, V1, V2
  3. V2, E, V1
  4. E, V2, V1
  Where E denotes the ETDRS assessment, V1 denotes the VDAP assessment in home environment 1, and V2 denotes the VDAP assessment in home environment 2.
  The randomization will be blocked in groups of 4 subjects to ensure balance for the VA testing sequences.
  Other Names: ETDRS Chart

SUMMARY:
Visual acuity is the relative ability of the eye to resolve detail that is usually expressed as the reciprocal of the minimum angular separation in minutes of two lines just resolvable as separate and that forms in the average human eye an angle of one minute.

Visibly Inc. has developed a method for determining a patient's visual acuity electronically via a web-based software system that can be self-administered wherever convenient. This method provides an efficient alternative for people to have immediate access to visual acuity measurements.

DETAILED DESCRIPTION:
The Visibly Digital Acuity Product (VDAP) is a web-based, self-guided software application intended for use by adults, ages 22 to 40, at home, to evaluate visual acuity with or without correction. The standalone software application allows the user to interface with the software via a web browser on two internet-enabled devices:

* A computer screen (the Display) which displays optotypes
* A touchscreen mobile device (the Remote) which operates as a remote control and interface for the user to respond to prompts related to the optotypes appearing on the Display while standing 10 feet away

The software allows users to view and respond to displayed optotypes and uses the responses to categorize a user's visual acuity into one of two buckets:

* 20/25 or better
* Worse than 20/25

ELIGIBILITY:
Inclusion Criteria:

* 1. Be between 22 and 40 years (inclusive) of age at the time of consent 2. Be able and willing to provide written informed consent, attend all scheduled visits and comply with all study procedures

Exclusion Criteria:

* 1. Have any of the following conditions (based on subject report):

  1. Advanced eye disease in either eye;
  2. Poor vision as a result of refractive surgery in either eye;
  3. Unable to walk;
  4. Unable to hear or follow audio instructions.

Ages: 22 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 358 (Actual)
Dates: Start 2021-07-22 (Actual); Primary Completion 2021-10-04 (Actual); Study Completion 2021-10-04 (Actual)

PRIMARY OUTCOMES:
Effectiveness | Up to 3 hours
  The proportion of study eyes with VDAP VA of 20/25 or better 20/25 or better [Positive Predictive Value (PPV)]
Reproducibility | Up to 3 hours
  The proportion of study eyes which receive the same VA classification (20/25 or Better vs. Worse than 20/25) for the two VDAP tests

SECONDARY OUTCOMES:
Effectiveness | Up to 3 hours
  The proportion of subjects with matching VDAP and ETDRS VA classifications (20/25 or Better vs. Worse than 20/25) for both eyes (study eye and non-study eye)
Reproducibility | Up to 3 hours
  The proportion of subjects with matching VDAP VA classifications (20/25 or Better vs. Worse than 20/25) for the two VDAP tests for both eyes (study eye and non-study eye)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Andover Eye Associates, Andover, Massachusetts
  - Core, Inc, Shelby, North Carolina
  - Total Eye Care, Memphis, Tennessee